CLINICAL TRIAL: NCT04467008
Title: Evaluation of Covid-19 Rapid Diagnostic Tests on Blood Drop
Brief Title: Covid-19 Rapid Diagnostic Tests on Blood Drop
Acronym: COVID-TEST
Status: Completed | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/05
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-07

CONDITIONS: Covid19
Keywords: Covid 19; Diagnostic; Biosynex; Blood drop
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One group of patients

SUMMARY:
This study will evaluate the diagnostic reliability of the Biosynex rapid blood test for Covid-19 infection.

DETAILED DESCRIPTION:
The Covid-19 pandemic requires a reliable diagnosis of affected patients in order to manage them in an appropriate manner, in the appropriate departments. Furthermore, the diagnostic reference at the time of this study is based on reverse transcription by reaction in polymerase chain reaction (RT-PCR) on a nasopharyngeal swab taken. This method has may yield false negatives (up to 30% depending on the series) and its lead time is several hours.

Alternatives are therefore being developed, in particular rapid blood tests. The rapid diagnostic test distributed by Biosynex has been evaluated by the National Reference Center for Respiratory Infections Viruses as very specific for the detection of IgG + IgM (93%).

As part of the evaluation of this test, it was used in patients with severe Covid-19 disease, requiring hospitalization in critical care in order to be able to establish their reliability in a clinical context where many confounding factors may occur, such as lymphopenia or systemic inflammation. However, the early diagnosis of this patient population remains critical in order to be able to refer them to the appropriate services.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 diagnosis with at least one positive RT-PCR

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed COVID-19 pneumonia (using RT-PCR) who required hospitalization in intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Positivity of the rapid diagnostic test | Immediate, up to 1 day.
  Positivity of the rapid diagnostic test, assessed by the presence of either IgM or IgG

CONTACTS AND LOCATIONS:
Overall Officials: Lee Nguyen, MD, Principal Investigator — CMC Ambroise Paré
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, France